CLINICAL TRIAL: NCT02030496
Title: Volar Internal Plate Fixation vs. Plaster in Extra- Articular Distal Radial Fractures
Acronym: VIPER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Onze Lieve Vrouwe Gasthuis (Other); Diakonessenhuis, Utrecht (Other); Elkerliek Hospital (Other); Groene Hart Ziekenhuis (Other); Dijklander Ziekenhuis (Other); Reinier de Graaf Groep (Other); Maasstad Hospital (Other); BovenIJ Hospital (Other); Rijnland Hospital (Other); Flevoziekenhuis (Other); Radboud University Medical Center (Other); Maxima Medical Center (Other); Zaans Medisch Centrum (Other)
Responsible Party: Principal Investigator, J.C. Goslings, Prof, PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL37754.018.12
Record Dates: First submitted 2014-01-06; First posted 2014-01-08 (Estimated); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Displaced Extra-articular Distal Radius Fractures
Keywords: distal radius fractures; Closed reduction; Open reduction internal fixation; Volar plate; Redislocation; Unstable fracture; Extra-articular fracture; Colles fracture; Barton fracture
MeSH Terms: conditions — Wrist Fractures; Colles' Fracture | interventions — Open Fracture Reduction; Fracture Fixation, Internal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Closed reduction and plaster (Active Comparator): Closed reduction will be performed and after adequate reduction has been confirmed, the wrist will be immobilised according to Dutch guidelines: a splint for one week followed by a circular cast for another four weeks.
  Interventions: Other: Closed reduction and plaster
- open reduction and internal fixation (Active Comparator): The intervention group will be treated with open reduction and internal fixation with a volar locking plate.
  Interventions: Procedure: open reduction and internal fixation

INTERVENTIONS:
Procedure: open reduction and internal fixation — The surgery will be performed by a certified trauma surgeon. After the fracture site is exposed, the fracture will be reduced and provisionally fixed with K-Wires and reduction forceps. An appropriate volar locking plate which best suits the anatomy of the wrist and the fracture type will be selected. Screw placement and fracture reduction will be confirmed intra-operatively by radiographic images. No post-operative fixation will be applied and patients will be instructed to use the affected extremity in daily activities as pain allows. According to Dutch treatment standards, vitamin C 500 milligrams will be prescribed to all patients at initial presentation and for a duration of two months in order to prevent Complex Regional Pain Syndrome.
  Arms: open reduction and internal fixation
Other: Closed reduction and plaster — Closed reduction will be performed according to the Robert-Jones method. This involves increasing the deformity first, then applying continuous traction and immobilising wrist and hand in the reduced position. Additional radiographs will be performed to verify the quality of the reduction. After this has been confirmed, the wrist will be immobilised according to Dutch guidelines: a splint for one week followed by a circular cast for another four weeks. According to Dutch treatment standards, vitamin C 500 milligrams will be prescribed to all patients at initial presentation and for a duration of two months in order to prevent Complex Regional Pain Syndrome.
  Arms: Closed reduction and plaster

SUMMARY:
BACKGROUND:

Fractures of the distal radius are common and account for an estimated 17% of all fractures diagnosed. Two-thirds of these fractures are displaced and require reduction. Although distal radius fractures are considered to be relatively harmless, inadequate treatment may result in impaired function of the wrist. The consequences of post-traumatic loss of function are comprehensive, both on an individual and a social level, and have long been underestimated. Despite the substantial implications, no evidence-based treatment method yet exists. Good results have been described both in patients treated conservatively and surgically. Nevertheless, 60% of all fractures redislocate after conservative treatment at which point surgical reduction and fixation is the treatment of choice. Recently, the use of volar locking plates has become more popular. This type of osteosynthesis employs a volar approach to the wrist and provides immediate stable fixation of the reduced fracture. This stability allows for early mobilisation and may therefore result in an improved regain of function. The aim of this study is to compare the functional outcome following surgical reduction and fixation with a volar locking plate with the functional outcome following closed reduction and plaster immobilisation at one year follow-up in patients with displaced extra-articular distal radius fractures.

DESIGN:

This single blinded randomised controlled trial will randomise between open reduction and internal fixation with a volar locking plate (intervention group) and closed reduction followed by plaster immobilisation (control group). The study population will consist of all consecutive adult patients who are diagnosed with a displaced extra-articular distal radius fracture which has been adequately reduced at the Emergency Department. The primary outcome (functional outcome) will be assessed by means of the Disability Arm Shoulder Hand Score (DASH). Since the treatment allocated involves a surgical procedure, randomisation status will not be blinded. However, the researcher assessing the outcome at one year will be unaware of the treatment allocation. In total, 90 patients will be included in this trial which will be conducted in the Academic Medical Centre Amsterdam and its partners of the regional trauma care network.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years and ≤ 75 years
* Extra-articular (AO type A) displaced distal radius fracture, as classified on lateral, posterior anterior and lateral carporadial radiographs by a radiologist or trauma surgeon.
* Acceptable closed reduction obtained according to current Dutch guidelines within 12 hours after presentation at the Emergency Department (ED).

Exclusion Criteria:

* Open distal radius fractures
* Multiple trauma patients (Injury Severity Score (ISS) ≥16)
* Other fractures of the affected extremity
* Patients with impaired wrist function prior to injury due to arthritis/neurological disorders of the upper limb
* Patient suffering from disorders of bone metabolism, connective tissue or (joint) hyperflexibility.
* Insufficient comprehension of the Dutch language to understand the treatment information and informed consent forms as judged by the attending physician.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Wrist function/pain/disability at one year assessed with DASH score | At12 months follow up
  the primary endpoint of this study is wrist function, pain and disability as measured with the DASH score. The Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire is a 30-item, self-report questionnaire designed to measure physical function and symptoms in patients with any or several musculoskeletal disorders of the upper limb.

SECONDARY OUTCOMES:
Wrist function at one year assessed with PRWE score | 6 weeks, three, six and 12 months
  The PRWE questionnaire is a 15-item questionnaire designed to measure wrist pain and disability in activities of daily living. The PRWE allows patients to rate their levels of wrist pain and disability from 0 to 10, and consists of three subscales: Pain, Function and Cosmetics.
Quality of Life | 6 weeks, three, six and 12 months
  Quality of Life assessed using the Short Form-36 (SF-36) questionnaire. The SF-36 is a validated multipurpose, short form health survey which contains 36 questions representing eight different health domains. These domains are combined into a mental and physical component scale. From each domain, scores ranging from 0 to 100 points are derived, with lower scores indicating poorer quality of life.
Pain | 6 weeks, 3, 6 and 12 months
  Pain as indicated on a visual Analogue Scale (VAS), in which 0 implies no pain and 10 the worst possible pain. Patients will be asked to give an estimation of the type and quantity of pain medication taken during all follow-up visits.
Patient satisfaction | at one year
  Patient satisfaction at one year by simply asking patients if they are satisfied with the result (yes/no).
Range of motion | 6 weeks, 3, 6 and 12 months
  Range of motion of the wrist measured on both sides with a handheld goniometer.
Grip strength | 6 weeks, 3, 6 and 12 months
  Grip strength as measured with a dynamometer.
Radiological parameters | At one year
  Radiological parameters: radial inclination, volar/dorsal tilt, comminution, ulnar variance and radial length measured digitally in the Picture Archiving and Communication System (PACS) on standard posterior anterior (PA), lateral carporadial and lateral X-rays of the wrist. Radiographs will be obtained according to standardised procedures. PA radiographs with the shoulder in 90 degrees abduction, elbow in 90 degrees flexion and the wrist in neutral position; lateral X-rays with the shoulder in neutral position and elbow in 90 degrees flexion; and the lateral carporadial radiographs will be obtained by positioning the lower arm on a 20-25 degrees angled wedge.
Complications | 1 week, 2-3 weeks, 6 weeks, 3, 6 and 12 months
  Complication rate such as: loss of reduction, cross-overs from conservative to operative treatment, fracture malunion or non-union, wound and/or plate infection, tendon irritation and/or rupture, neuropathy and the occurrence of complex regional pain syndrome.

CONTACTS AND LOCATIONS:
Overall Officials: J. Carel Goslings, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, Amsterdam, Netherlands